CLINICAL TRIAL: NCT03336892
Title: Mental Health Care Coordination for Transition Aged Youth With Serious Emotional Disturbance/Serious Mental Illness
Brief Title: Mental Health Care Coordination for Transition Aged Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Tuchman, Principal Investigator, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro7512; R40MC29453 (Other Grant/Funding Number: HRSA Maternal and Child Health Bureau)
Record Dates: First submitted 2017-10-23; First posted 2017-11-08 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Mental Health
Keywords: Care Coordination
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enhanced usual care with written mental health resources and system navigation information in addition to individualized mental health care coordination by a dedicated specially trained mental health care coordinator.
  Interventions: Behavioral: Mental Health Care Coordination
- Control (No Intervention): Enhanced usual care with written mental health resources and system navigation information.

INTERVENTIONS:
Behavioral: Mental Health Care Coordination — Enhanced usual care with written mental health resources and system navigation information in addition to individualized mental health care coordination by a dedicated specially trained mental health care coordinator.
  Arms: Intervention

SUMMARY:
This study seeks to quantify the impact of recommended mental health care coordination practices on patient experiences of care, (i.e. satisfaction, stigma, quality of mental health care), evaluate the efficiency and effectiveness of the intervention (i.e. care coordination, timing, unmet needs), and assess mental health outcomes (i.e. symptoms and functioning, involvement with law enforcement/juvenile justice system; rates of substance use /abuse, service utilization) in a population of 16-22 year-old youth receiving primary care in a D.C. urban academic adolescent medicine practice, using standardized outcome measures.

DETAILED DESCRIPTION:
In the maternal and child health field, there is increasing awareness of modifiable health conditions that appear early in the life course and impact development and wellness throughout the life span. Special opportunities exist in vulnerable populations with serious mental health conditions to better understand what life course events can facilitate attainment of optimal health and development. One such opportunity is making sure youth with serious emotional disturbance/serious mental illness receive the mental health services they need.

Unfortunately, untreated mental illness among adolescents and young adults is a major public health problem. Particularly concerning is the fact that 80% of youth with serious emotional disturbance/serious mental illness are not receiving needed mental health services and unmet mental health needs are even higher among certain populations, including minority youth. Youth with untreated mental health problems face a number of challenges that are exacerbated when left untreated. For example, youth with serious mental illness tend to have more difficulties in school and more involvement with the criminal justice system than their peers. These youth also face more challenges successfully transitioning to adulthood and becoming productive members of society.

Untreated mental illness tends to lead to more intensive and costly treatment down the road. There are many barriers to accessing mental health services, including stigma and difficulty navigating a complex mental health system, which contribute to unmet mental health needs. Additionally, youth may be so significantly impaired that expecting them to access mental treatment without some supportive services is unrealistic.

In light of these facts, it becomes urgent to implement recommended standards for mental health integration and evaluate their impact on mental health outcomes. The Center for Integrated Health Solutions in a joint Health Resources and Services Administration (HRSA)-Substance Abuse and Mental Health Services Administration (SAMHSA) effort recently released expanded joint principles for behavioral health integration. In this model, coordinated care is defined by primary and behavioral health care provided at different locations in the medical neighborhood, but care is coordinated through enhanced communication across the two disciplines. This report makes available an important standard for establishing integrated mental health care coordination practices within a primary care setting, but also demands careful evaluation.

This study seeks to quantify the impact of recommended mental health care coordination practices on patient experiences of care, (i.e. satisfaction, stigma, quality of mental health care), evaluate the efficiency/effectiveness of the intervention (i.e. care coordination, timing, unmet needs), and assess mental health outcomes (i.e. symptoms and functioning, involvement with law enforcement/juvenile justice system; rates of substance use /abuse, service utilization) in a population of 16-22 year-old youth receiving primary care in a D.C. urban academic adolescent medicine practice, using standardized outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* has a diagnosis of serious emotional disturbance/serious mental illness
* has not received outpatient mental health services in the past 30 days

Exclusion Criteria:

* does not have a diagnosis of serious emotional disturbance/serious mental illness
* has received outpatient mental health services in the past 30 days

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Connection to mental healthcare | 2 years
  Number of study participants self-reported receiving mental health care services since enrollment

SECONDARY OUTCOMES:
Patient Experiences | 2 years
  Experience of Care and Health Outcomes (ECHO) Survey
Depression symptoms | 2 years
  PHQ-9 Questionnaire
Mental Health Stigma | 2 years
  Internalized Stigma of Mental Illness (ISMI) Questionnaire
Patterns of substance use | 2 years
  Youth Risk Behavior Survey (YRBS) Questionnaire
Adverse Childhood Events | 2 years
  Philadelphia ACE Survey

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Tuchman, MD, MPH, Principal Investigator — Children's National Research Institute